CLINICAL TRIAL: NCT07062263
Title: Trastuzumab Plus Chemotherapy vs Chemotherapy Alone in First-line HER2 Positive Advanced Biliary Tract Cancer Patients - a Randomized Non-blinded Two-arm Phase III Prospective Clinical Trial (TAB-2 Study).
Brief Title: Trastuzumab Plus Chemotherapy vs Chemotherapy Alone in First-line HER2 Positive Advanced Biliary Tract Cancer Patients
Acronym: TAB-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr. Vikas Ostwal, Professor Dept of Medical Oncology, Convener Gastro-Intestinal Disease Management Group, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4172
Record Dates: First submitted 2025-06-30; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Biliary Tract Cancer; HER2-positive Cancer; Advanced Cancer; Unresectable Biliary Tract Carcinoma; Metastatic Biliary Tract Carcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Trastuzumab; Drug Therapy; Gemcitabine; Cisplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Phase III open-label parallel design randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Trastuzumab plus Chemotherapy (Experimental): Trastuzumab + Gemcitabine + cisplatin
  * Gemcitabine 1000 mg/m2 IV over 30 mins on day 1 and day 8 q 3 weekly
  * Cisplatin 25 mg/m2 IV over 60 minutes on day 1 and day 8 q 3 weekly
  * Trastuzumab 8mg/kg IV over 90 mins as first dose and subsequent doses at 6mg/kg IV over 30-60 minutes q 3 weekly (=1 cycle)
  OR
  * Trastuzumab with Gemcitabine-cisplatin-Nab-Paclitaxel
  * Gemcitabine 800 mg/m2 IV over 30 mins on day 1 and day 8 q 3 weekly
  * Nab-paclitaxel 100 mg/m2 IV over 1-2 hours on day 1 and day 8 q 3 weekly
  * Cisplatin 25 mg/m2 IV over 60 minutes on day 1 and day 8 q 3 weekly
  * Trastuzumab 8mg/kg IV over 90 mins as first dose and subsequent doses at 6mg/kg IV over 30-60 minutes q 3 weekly (=1 cycle) Start of next cycle on D22 Immunotherapy is allowed as per the discretion of the treating physician
  Interventions: Drug: Trastuzumab; Drug: Chemotherapy
- Arm B: Chemotherapy alone (Active Comparator): Gemcitabine + cisplatin
  * Gemcitabine 1000 mg/m2 IV over 30 mins on day 1 and day 8 q 3 weekly
  * Cisplatin 25 mg/m2 IV over 60 minutes on day 1 and day 8 q 3 weekly (=1 cycle)
  OR
  * Gemcitabine-cisplatin-Nab-Paclitaxel
  * Gemcitabine 800 mg/m2 IV over 30 mins on day 1 and day 8 q 3 weekly
  * Nab-paclitaxel 100 mg/m2 IV over 1-2 hours on day 1 and day 8 q 3 weekly =Cisplatin 25 mg/m2 IV over 60 minutes on day 1 and day 8 q 3 weekly (=1 cycle) Start of next cycle on D22 Immunotherapy is allowed as per the discretion of the treating physician
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Trastuzumab — Inj Trastuzumab given in a dose of 8mg/kg intravenously over 90 mins as first dose and subsequent doses at a dose of 6mg/kg intravenously over 30-60 minutes in 3 weekly cycle along with standard of care chemotherapy
  Other Names: Transtuzumab with standand of chemotherapy
  Arms: Arm A: Trastuzumab plus Chemotherapy
Drug: Chemotherapy — Gemcitabine + cisplatin OR Gemcitabine-cisplatin-Nab-Paclitaxel given as a standard of care, chemotherapy as per the institutional guidlines
  Other Names: Standard of chemotherapy; Gemcitabine; cisplatin; Nab-Paclitaxel

SUMMARY:
This is a randomized, open-label, two-arm, Phase III clinical trial evaluating the efficacy and safety of trastuzumab plus chemotherapy versus chemotherapy alone as first-line treatment in patients with HER2-positive advanced or metastatic biliary tract cancers (BTC). HER2-positive BTCs represent a molecular subset of these rare cancers, associated with poor prognosis and limited treatment options.

Eligible patients with histologically confirmed HER2-positive (IHC 3+ or IHC 2+ with FISH amplification) unresectable or metastatic biliary tract adenocarcinoma-including gallbladder cancer, intrahepatic, and perihilar cholangiocarcinoma-will be randomized in a 1:1 ratio. Participants in the intervention arm (Arm A) will receive either gemcitabine and cisplatin with or without nab-paclitaxel plus trastuzumab, while those in the control arm (Arm B) will receive chemotherapy alone (gemcitabine + cisplatin with or without nab-paclitaxel). Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, or death.

The primary endpoint is 6-month progression-free survival (PFS). Secondary endpoints include overall survival (OS), response rate (RR), quality of life (QOL), and adverse event (AE) profiles. The study aims to enroll 196 patients across a single center in India over a period of 5 years, with an additional 6-month follow-up. This trial builds on earlier Phase II findings suggesting improved outcomes with trastuzumab in HER2-positive BTC and aims to provide the first randomized evidence for the benefit of HER2-targeted therapy in this setting.

DETAILED DESCRIPTION:
Title of study- Trastuzumab plus chemotherapy vs Chemotherapy alone in first-line HER2 positive advanced biliary tract cancer patients - a randomized non-blinded two-arm Phase III prospective clinical trial (TAB - 2 study)

Indication- HER2-positive advanced/metastatic biliary tract cancers fit for first-line chemotherapy with gemcitabine-based combination

Type of Study- Two arm open-label prospective Phase III parallel design randomized superiority clinical trial

Biliary tract cancers (BTC), including gallbladder cancer and cholangiocarcinomas, are uncommon but aggressive tumors with poor prognosis in the advanced or metastatic setting. The current standard first-line treatment is gemcitabine combined with a platinum agent, which offers limited benefit. Emerging molecular profiling has identified HER2 overexpression or amplification in a subset of BTCs, particularly in gallbladder cancer, and has opened new avenues for targeted therapy.

Trastuzumab, a monoclonal antibody targeting the HER2 receptor, has shown clinical activity in HER2-positive BTCs in early-phase studies. Preliminary evidence from a single-arm Phase II study (TAB trial) suggests that combining trastuzumab with chemotherapy may significantly improve progression-free survival in treatment-naïve HER2-positive patients.

The TAB-2 study is a prospective, randomized, open-label Phase III trial designed to evaluate whether adding trastuzumab to first-line chemotherapy improves clinical outcomes in patients with HER2-positive advanced BTC. Patients will be randomized to receive chemotherapy with or without trastuzumab. Chemotherapy regimens may include gemcitabine and cisplatin, with or without nab-paclitaxel, based on physician discretion. Trastuzumab will be administered every three weeks along with chemotherapy until disease progression, unacceptable toxicity, or withdrawal of consent.

The study will be conducted at a single academic center in India, with a planned enrollment of 196 participants over 5 years. This trial aims to provide definitive randomized evidence regarding the benefit of incorporating HER2-targeted therapy into the first-line treatment of advanced BTC and to inform future clinical practice for this rare molecular subtype.

Primary endpoint- To evaluate the difference in progression-free survival (PFS) at 6 months between Trastuzumab - chemotherapy combination and chemotherapy alone.

Treatment scheme

1. Arm A (Trastuzumab plus chemotherapy)-Gemcitabine plus Trastuzumab OR Gemcitabine Plus Cisplatin Plus Nab-paclitaxel on D1 and D8 Plus Trastuzumab D1 Start of next cycle on D 22
2. Arm B (Chemotherapy alone)- Gemcitabine Plus Cisplatin D1 and D8 q 21 days OR Gemcitabine Plus Cisplatin Plus Nab-paclitaxel D1 and D8) Start of next cycle on D 22 Treatment in both arms will be continued till unacceptable toxicity, death, or consent withdrawal.

In both arms Immunotherapy is allowed as per the discretion of the treating physician

Sample Size calculation- Based published phase 2 single-arm TAB trial, the median PFS in HER2 positive biliary tract cancer with Trastuzumab plus chemotherapy was approximately 8 months (6-month PFS was approximately 75 - 80%), while the median PFS with chemotherapy alone ranges from 5-6 months (6-month PFS approximately 55%-65%). Assuming the Trastuzumab combination will increase the 6-month PFS to 75% in comparison to 55% with chemotherapy alone, with a power of 80% and alpha of 0.05 and margin of risk difference of 3 %, a Phase III randomized study will require a total of 196 patients (98 per arm), assuming an attrition rate of 5 % per arm with a study accrual period of 5 years. Follow up the duration of the study will be 6 months post-accrual of the last patient.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed adenocarcinoma of the biliary tract, with the following specifications -

1. Biliary tract cancers include gallbladder cancer, intrahepatic cholangiocarcinoma, and perihilar cholangiocarcinoma.
2. HER2-positive by IHC or FISH
3. Age >=18 years.
4. ECOG performance status 0 - 2.
5. Unresectable or metastatic cancer.
6. Patient does not have any contraindications to receive chemotherapy or trastuzumab.
7. Adequate hematological, hepatic, and renal function parameters- Hematological- Hb> 80 g/L, ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L. Liver functions- bilirubin ≤ 2 x upper limit normal (ULN), AST/ALT ≤ 5 x ULN, alkaline phosphatase ≤ 6 x upper limit normal (ULN) S. albumin ≥ 30 g/L.

   Renal function- Creatinine ≤ 1.5 ULN, Creatinine clearance >= 30 mL/min.
8. Normal cardiac ejection fraction and cardiac function, as assessed by echocardiography, ejection fraction (EF) >=50% or above the lower limit of normal. ECG with no clinically relevant abnormalities.
9. Women of childbearing age should have a negative pregnancy test at the time of randomization and should be willing to use adequate contraception during the treatment phase of the trial.
10. Subjects must provide written informed consent prior to the performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up assessments and procedures.
11. Subjects who have received adjuvant chemotherapy will be considered eligible provided that therapy is completed more than 12 months before study enrollment. Patients who have received radiation therapy and surgery will also be eligible provided the interventions have been completed 3 and 2 weeks, respectively, before enrolment in the study.
12. Negative serum pregnancy test (if applicable) and willing for adequate contraception.
13. At least one measurable disease according to RECIST criteria.
14. Life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Distal cholangiocarcinoma
2. Known hypersensitivity or contraindications against gemcitabine, cisplatin, Nab- paclitaxel, or trastuzumab.
3. Clinically significant active coronary heart disease, cardiomyopathy, or congestive heart failure, NYHA III-IV.
4. Clinically significant valvular defect.
5. Past or current history of other malignancies not curatively treated and without evidence of disease for more than 5 years, except for curatively treated basal cell carcinoma of the skin and in situ carcinoma of the cervix.
6. Severe dyspnea at rest due to complications of advanced malignancy or requiring supplementary oxygen therapy.
7. Baseline neuropathy > NCI Grade I.
8. Subject pregnant or breastfeeding, or planning to become pregnant within 6 months after the end of treatment.
9. Received prior chemotherapy within 1 year.
10. Any active ILD/ history of lung illness requiring bronchodilator drugs.
11. Patients with prior chemotherapy for metastatic disease will be ineligible for enrollment in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | at 6 month after randomisation
  the time from the time of diagnosis of an advanced disease to the time of disease progression or loss to follow-up or death, whichever is earlier

SECONDARY OUTCOMES:
Overall survival (OS) | at 6month, 1 year from the date of randomisation or till the time of death, lost to follow-up or last observation, whichever is earlier
  the time from the time of diagnosis to the time of death, lost to follow-up or last observation, whichever is earlier
Response rates | at 6th month from the date of randomisation
  measured as per RECIST criteria in CE CT scan as compare with the baseline scans
Quality of life (QOL) | at baseline and at completion of 4 cycles of chemotherapy (each cycle is 22 days)
  measured using the EORTC-QLQ-30 questionnaires All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level
Safety profile | "At the end of each Cycle (each cycle is 22 days)
  side effects and adverse event profile with the combination will be reported as NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Ostwal, DM, Principal Investigator — Tata Memorial Hospital, Parel, Mumbai, Maharashtra, India 400012
Locations (6):
- India (6):
  - Homi Bhabha Cancer Hospital and Research Centre, Muzaffarpur, Muzaffarpur, Bihar
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Institute of Medical Sciences & SUM Hospital, Bhubaneswar, Odisha
  - Homi Bhabha Cancer Hospital and Research Centre, Mūllānpur, Punjab
  - Mahamana Pandit Madan Mohan Malviya Cancer Centre (MPMMC) and Homi Bhabha Cancer Hospital (HBCH), Varanasi, Uttar Pradesh
  - MAX Super Speciality Hospital, SAKET, Delhi

IPD SHARING:
Plan to Share IPD: No